CLINICAL TRIAL: NCT00003542
Title: Phase I/II Study of Subcutaneous Administration of Pegylated-Interferon Alpha-2A (RO 25-8310) in Previously Untreated Patients With Locally Advanced or Metastatic Renal Cell Carcinoma
Brief Title: Interferon Alfa in Treating Patients With Advanced Kidney Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 98-052; CDR0000066596 (Registry Identifier: PDQ (Physician Data Query)); ROCHE-NO15753C; UCLA-9903045; NCI-G98-1475
Record Dates: First submitted 1999-11-01; First posted 2004-08-04 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Kidney Cancer
Keywords: stage III renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell

INTERVENTIONS:
Biological: pegylated interferon alfa

SUMMARY:
RATIONALE: Interferon alfa may interfere with the growth of cancer cells.

PURPOSE: Phase I/II trial to study the effectiveness of interferon alfa in treating patients with advanced kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose (MTD) of pegylated-interferon alfa-2a in patients with advanced or metastatic renal cell carcinoma. II. Evaluate the safety profile of the MTD in this patient population. III. Determine the objective response rate, time to response, duration of response, time to progression, and survival rate in this patient population.

OUTLINE: This is a dose escalation, open label, multicenter study. Patients receive pegylated-interferon alfa-2a (PEG-IFN) subcutaneously once a week for 24 weeks. Dose escalation of PEG-IFN continues until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity. After the MTD of PEG-IFN is determined, additional patients are treated at this dose level. These patients may continue treatment after the first 24 weeks for up to 1 year, in the absence of disease progression. Patients are followed for 4 weeks.

PROJECTED ACCRUAL: A total of 46-58 patients will be accrued for this study within 9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed advanced or metastatic renal cell carcinoma Bidimensionally measurable lesions that have not been irradiated Minimum indicator lesion size: Liver, soft tissue, or other masses - one diameter at least 20 mm (evaluable only radiographically) Lung - one diameter at least 10 mm by x-ray or CT scan Skin lesions and lymph nodes - one diameter at least 10 mm by clinical measurement No clinical or radiologic evidence of CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 80-100% Life expectancy: Not specified Hematopoietic: WBC at least 3000/mm3 Neutrophil count at least 1500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10 g/dL (red cell transfusions allowed) Hepatic: Bilirubin no greater than 1.5 times the upper limit of normal (ULN) (except for patients with Gilbert's syndrome) ALT and/or AST no greater than 2.5 times ULN (no greater than 4 times ULN with liver metastases) Alkaline phosphatase no greater than 2.5 times ULN (no greater than 4 times ULN with liver metastases) Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No history of severe cardiac disease: New York Heart Association class II (if not due to cancer), III, or IV Myocardial infarction within the past 6 months Ventricular tachyarrhythmias requiring ongoing treatment Unstable angina Other: Not pregnant or nursing Fertile patients must use effective contraception No other prior or concurrent malignancy except basal cell carcinoma of the skin, carcinoma in situ of the cervix, or any other malignancy from which the patient has been disease free for at least 2 years No history of medically significant psychiatric disease, especially depression No history or evidence of retinopathy No seizure disorders

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior or concurrent immunotherapy, biologic response modifiers, cytokines, monoclonal antibodies, antitumor vaccines, or any other systemic therapy Chemotherapy: No prior or concurrent chemotherapy Endocrine therapy: No prior or concurrent hormone therapy Hormone replacement after adrenalectomy is allowed Radiotherapy: Prior radiotherapy allowed No concurrent radiotherapy Surgery: Prior nephrectomy allowed Other: No other concurrent investigational drugs No concurrent anticonvulsant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 1998-05; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Motzer, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Memorial Sloan-Kettering Cancer Center, New York, New York